CLINICAL TRIAL: NCT03378375
Title: Resting Energy Expenditure Equations in Amyotrophic Lateral Sclerosis, Creation of a ALS-specific Equation
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: ALS/jesus
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nutritional assessement

SUMMARY:
Introduction: Resting energy expenditure (REE) formulas for healthy people (HP) are used to calculate REE (cREE) in amyotrophic lateral sclerosis (ALS) patients. In ALS an increase of measured REE (mREE) in indirect calometry (IC) compared to cREE is found in 50-60%. The aims were (i) to assess accuracy of cREE assessed using eleven formulas as compared to mREE and (ii) to create if needed a specific cREE formula for ALS patients.

Method: ALS patients followed in the ALS expert center of Limoges between 1996 and 2014 and with a nutritional evaluation were included. mREE assessed with IC and cREE calculated with eleven predictive formulas (Harris Benedict (HB) 1919, HB 1984, WSchofield, De Lorenzo, Johnstone, Mifflin, WHO/FAO, Owen, Fleisch, Wang and Rosenbaum) were collected at time of diagnosis. Fat free mass (FFM) and fat mass (FM) were measured with impedancemetry. A Bland and Altman analysis was carried out. The percentage of accurate prediction ± 10%of mREE, and intraclass correlation coefficients (ICC) were calculated. Using a derivation sample, a new REE formula was created using multiple linear regression according to sex, age, FFM and FM. Accuracy of this formula was assessed in a validation sample.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosed patients according to Airlie House criteria
* treated with riluzole
* respiratory quotient (RQ) of patients in indirect calorimetry (IC) should be in between 0.7 and 0.87

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS diagnosed patients according to Airlie House criteria
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 1996-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure emeasures | nutritional assessement should have been be performed within a 1.5 months' time period. IC had to be performed no later than 12 months after diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU LImoges, Limoges, France